CLINICAL TRIAL: NCT04895735
Title: Phase II Study of Pemetrexed and Pembrolizumab in Recurrent and/or Metastatic Salivary Gland Malignancies
Brief Title: MC200708 Pemetrexed and Pembrolizumab for the Treatment of Recurrent and/or Metastatic Salivary Gland Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC200708; NCI-2021-04161 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20-010144 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2021-05-18; First posted 2021-05-20 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Salivary Gland Carcinoma; Recurrent Salivary Gland Carcinoma; Stage IV Major Salivary Gland Cancer AJCC v8; Adenoid Cystic Carcinoma
MeSH Terms: conditions — Salivary Gland Neoplasms; Carcinoma, Adenoid Cystic | interventions — pembrolizumab; Pemetrexed; Specimen Handling; Magnetic Resonance Spectroscopy; Glutamate Carboxypeptidase II

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab, pemetrexed) (Experimental): Patients receive pembrolizumab IV over 30 minutes and pemetrexed disodium IV over 10 minutes on day 1. Treatment with pembrolizumab repeats every 21 days for up to 35 cycles (2 years) in the absence of disease progression or unacceptable toxicity. Cycles of pemetrexed disodium repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients who had stable disease, partial response, or complete response after completion of 35 cycles of pembrolizumab, may continue pembrolizumab for an additional 17 cycles (1 year) in the absence of disease progression or unacceptable toxicity. Patients additionally undergo blood sample collection, CT, PET/CT or MRI and may also undergo PSMA PET on study.
  Interventions: Biological: Pembrolizumab; Drug: Pemetrexed Disodium; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Procedure: Magnetic Resonance Imaging; Procedure: PSMA PET Scan

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Drug: Pemetrexed Disodium — Given IV
  Other Names: Alimta; Almita; LY231514; N-[4-[2-(2-Amino-4,7-dihydro-4-oxo-1H-pyrrolo[2,3-d]pyrimidin-5-yl)ethyl]benzoyl]-L-glutamic Acid Disodium Salt
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; Computerized axial tomography (procedure); Computerized Tomography (CT) scan; tomography
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; nuclear magnetic resonance imaging; sMRI; Structural MRI
Procedure: PSMA PET Scan — Undergo PSMA PET
  Other Names: Prostate-specific Membrane Antigen PET; PSMA PET; PSMA-Positron emission tomography

SUMMARY:
This phase II trial studies the effect of pemetrexed and pembrolizumab in treating patients with salivary gland cancer that has come back (recurrent) and/or has spread to other places in the body (metastatic). Chemotherapy drugs, such as pemetrexed, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. The purpose of this study is to evaluate whether pembrolizumab, an immunotherapy drug, in combination with the chemotherapy drug, pemetrexed, has an effect on advanced salivary gland cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the clinical benefit rate (CBR) of the combination of pembrolizumab and pemetrexed in patients with recurrent or metastatic adenoid cystic salivary gland cancer. (Group A1, adenoid cystic carcinoma [ACC]) II. To determine the response rate of the combination of pembrolizumab and pemetrexed in patients with recurrent or metastatic salivary gland cancer (recurrent/metastatic salivary gland cancer [R/M SGC]). (Groups A and B, ACC and non-ACC)

SECONDARY OBJECTIVES:

I. To determine the progression-free survival (PFS), overall survival (OS), response rate (ACC cohort), CBR rate (non-ACC), and adverse events of the combination of pembrolizumab and pemetrexed in patients with recurrent or metastatic salivary gland cancer (R/M SGC).

II. To assess safety and tolerability of the combination of pembrolizumab and pemetrexed in patients with recurrent or metastatic salivary gland cancer (R/M SGC).

CORRELATIVE RESEARCH OBJECTIVES:

I. To investigate the frequency of MTAP loss by immunohistochemistry in R/M SGC and whether it correlates with enhanced response to pemetrexed.

II. To measure the degree of PDL1 expression using formalin-fixed tumor samples, and determine the extent of PDL1 expression correlates with response to study treatment.

III. To investigate expression of thymidylate synthase by immunohistochemistry in R/M SGC and whether it correlates with enhanced response to pemetrexed.

IV. To investigate circulating tumor deoxyribonucleic acid (DNA) (ctDNA) and correlation with response to study treatment.

V. To prospectively investigate circulating prostate-specific membrane antigen (PSMA) extracellular vesibles (EVs) and correlate with disease burden and treatment response for patients with adenoid cystic carcinoma in Cohort A1.

VI. To prospectively investigate PSMA positron emission tomography (PET)/computed tomography (CT) as an imaging modality for patients with adenoid cystic carcinoma in Cohort A1.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes and pemetrexed disodium IV over 10 minutes on day 1. Treatment with pembrolizumab repeats every 21 days for up to 35 cycles (2 years) in the absence of disease progression or unacceptable toxicity. Cycles of pemetrexed disodium repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients who had stable disease, partial response, or complete response after completion of 35 cycles of pembrolizumab, may continue pembrolizumab for an additional 17 cycles (1 year) in the absence of disease progression or unacceptable toxicity. Patients additionally undergo blood sample collection, CT, PET/CT or magnetic resonance imaging (MRI) and may also undergo PSMA PET on study.

After completion of study intervention, patients are followed up at 30 days, and then every 3 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* REGISTRATION - INCLUSION CRITERIA
* Age >= 18 years
* Histologically confirmed diagnosis of recurrent or metastatic salivary gland cancer not amenable to curative-intent therapy
* COHORT A1: Rochester Minnesota only: Diagnosis of adenoid cystic carcinoma (ACC)
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 criteria

  * NOTE: Tumor lesions in a previously irradiated area are considered measurable disease if progression has been demonstrated in such lesions. Disease that is measurable by physical examination only is not eligible
* Prior treatment:

  * Prior treatment with checkpoint inhibitor(s) allowed
  * Any number of lines of prior therapy in the recurrent/metastatic setting is permitted at the investigator's discretion
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1

  * NOTE: PS must be assessed again within 7 days prior to first dose of study drug
* Hemoglobin >= 9.0 g/dL (obtained =< 8 days prior to registration)

  * NOTE: Must be met without growth factor support and no transfusions <14 days prior to testing
* Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 8 days prior to registration)
* Platelet count >= 100,000/mm^3 (obtained =< 8 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (obtained =< 8 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) =< 2.5 x ULN (=< 5 x ULN for patients with liver involvement) (obtained =< 8 days prior to registration)
* Prothrombin time (PT)/international normalized ratio (INR)/activated partial thromboplastin time (aPTT) =< 1.5 x ULN OR if patient is receiving anticoagulant therapy and INR or aPTT is within target range of therapy (obtained =< 8 days prior to registration)
* Creatinine =< 1.5 x ULN OR calculated creatinine clearance >= 45 ml/min using the Cockcroft-Gault formula (obtained =< 8 days prior to registration)
* Negative pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only

  * Note: If testing done for eligibility is > 72 hours prior to first dose, then pregnancy testing must be repeated and result must be negative for patient to receive treatment
* Persons able to become pregnant OR able to father a child must be willing to use an adequate method of contraception while on treatment and for 180 days after last treatment
* Life expectancy >= 12 weeks
* Provide written informed consent
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Willingness to provide mandatory blood specimens for correlative research
* Willingness to provide mandatory tissue specimens for correlative research

Exclusion Criteria:

* REGISTRATION - EXCLUSION CRITERIA
* Any of the following because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential and persons able to father a child who are unwilling to employ adequate contraception
  * Persons expecting to conceive or father children during study treatment or within 180 days (6 months) after the last treatment
* Any of the following prior therapies:

  * Surgery < 3 weeks prior to registration
  * Systemic anti-cancer therapy < 3weeks prior to registration
  * Radiotherapy < 2 weeks prior to registration OR Palliative radiation < 1 week prior to registration

    * NOTES: Must have recovered from all radiation related adverse effects (=< grade 1) Must not currently require corticosteroids Must not have had radiation pneumonitis
  * Live vaccine < 4 weeks prior to registration

    * NOTES: Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist) are live attenuated vaccines and are not allowed
  * Received an investigational agent or used an investigational device or participated in a study of an investigational agent < 4 weeks prior to registration
* Known active human immunodeficiency virus (HIV) infection (defined as patients who are not on anti-retroviral treatment and have detectable viral load and CD4+ < 500/ml)

  * NOTE: HIV-positive patients who are well controlled on anti-retroviral therapy are allowed to enroll
* Active autoimmune disease requiring systemic treatment < 2 years prior to registration, documented history of severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents with use of disease modifying agents, corticosteroids or immunosuppressive drugs

  * NOTE: Exceptions are allowed for:

    * Vitiligo
    * Resolved childhood asthma/atopy
    * Intermittent use of bronchodilators or inhaled steroids
    * Daily steroids at dose of =< 10 mg of prednisone (or equivalent)
    * Local steroid injections
    * Stable hypothyroidism on replacement therapy
    * Stable diabetes mellitus on therapy (with or without insulin)
    * Sjogren's syndrome
    * Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed
* Current or prior use of immunosuppressive medication < 14 days prior to registration

  * NOTE: The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intraarticular injection)
    * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent

      * Steroids as premedication for hypersensitivity reactions (e.g., premedication for computed tomography [CT] scans)
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection requiring systemic therapy
  * Interstitial lung disease or clinically significant pleural effusion
  * Clinically significant ascites
  * Serious, chronic gastrointestinal conditions associated with diarrhea (e.g., Crohn's disease or others)
  * Known history of hepatitis B (i.e., known positive hepatitis B virus [HBV] surface antigen [HBsAg] reactive)
  * Known active hepatitis C (i.e., positive for hepatitis C virus [HCV] ribonucleic acid [RNA] detected by polymerase chain reaction [PCR])
  * Known active tuberculosis (TB)
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Unstable cardiac arrhythmia or
  * Psychiatric illness/social situations that would limit compliance with study requirements (e.g., substance abuse)
* Co-morbid systemic illnesses or other severe concurrent disease or current evidence of any condition, therapy, or laboratory abnormality which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Failure to recover to =< grade 1 (or baseline) from adverse events due to previously administered therapies or prior surgery

  * Exceptions: Neuropathy, fatigue, and/or alopecia may be grade 1
* Known active central nervous system (CNS) metastases

  * NOTE: Patients with previously treated brain metastases may participate provided all of the following are true:

    * They are stable (without evidence of progression by imaging =< 4 weeks prior to registration and any neurologic symptoms have returned to baseline)
    * Have no evidence of new or enlarging brain metastases, and
    * Are not using steroids =< 14 days prior to registration
* Known leptomeningeal disease
* Hypersensitivity (>= grade 3) to pembrolizumab or any of its excipients
* Previous serious adverse event (>= grade 3) attributed to prior checkpoint inhibitor therapy
* History of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* History of grade >= 3 immune-related adverse event or any grade of immune-related neurologic or ocular adverse event while receiving immunotherapy

  * Note: Patients who had endocrine adverse events =< grade 2 are allowed to enroll if they are stable on appropriate replacement therapy and asymptomatic
* Other active malignancy < 2 years prior to registration

  * EXCEPTIONS: Non-melanotic skin cancer, superficial bladder cancer, papillary thyroid cancer, or carcinoma-in-situ of the cervix or others curatively treated and now considered to be at less than 30% risk of relapse
* History of allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2025-08-13 (Actual); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Confirmed response rate | Up to 24 weeks
  Evaluated by Response Evaluation Criteria in Solid Tumors version 1.1.
Clinical benefit rate (CBR) | Up to 24 weeks
  CBR will be defined as the rate of patients with stable disease, partial response or complete response as their best response during treatment.

SECONDARY OUTCOMES:
Overall survival | From study entry to death from any cause, assessed up to 3 years
  Estimated using the Kaplan-Meier method.
Progression-free survival | From study entry to the first of either disease progression or death from any cause, assessed up to 3 years
  Estimated using the Kaplan-Meier method.
Incidence of adverse events | Up to 3 years
  The maximum grade for each type of adverse event will be summarized using Common Terminology Criteria for Adverse Events version 5.0. The frequency and percentage of grade 3+ adverse events will be estimated.
Response rate [adenoid cystic carcinoma (ACC) cohort] | Up to 3 years
  Response rate will be assessed using RECIST 1.1 criteria. The data will be reported descriptively, with frequencies and percentages.
CBR (non-ACC cohort) | Up to 3 years
  CBR will be reported descriptively, with frequencies and percentages.

OTHER OUTCOMES:
Frequency of MTAP loss | Up to 3 years
  Assessed by immunohistochemistry. Will investigate correlation with enhanced response to pemetrexed. The associations of these markers with response will be done via Chi-square or Fisher's exact tests by cohort for categorical biomarkers and done via 2-sample t-tests (or the Wilcoxon Rank-Sum test) by cohort for continuous biomarker data. Descriptive statistics and tables will be reported.
Degree of PDL1 expression using formalin-fixed tumor samples | Up to 3 years
  Will determine the extent of PDL1 expression correlation with response to study treatment. The associations of these markers with response will be done via Chi-square or Fisher's exact tests by cohort for categorical biomarkers and done via 2-sample t-tests (or the Wilcoxon Rank-Sum test) by cohort for continuous biomarker data. Descriptive statistics and tables will be reported.
Expression of thymidylate synthase | Up to 3 years
  Assessed by immunohistochemistry. Will investigate correlation with enhanced response to pemetrexed. The associations of these markers with response will be done via Chi-square or Fisher's exact tests by cohort for categorical biomarkers and done via 2-sample t-tests (or the Wilcoxon Rank-Sum test) by cohort for continuous biomarker data. Descriptive statistics and tables will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A. Price, MD, Principal Investigator — Mayo Clinic in Rochester; Ashish Chintakuntlawar, MBBS, PhD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials